CLINICAL TRIAL: NCT00226551
Title: ß2 Adrenergic Receptor Polymorphisms and Vasodilation of Internal Mammary Artery Induced by Isoproterenol
Brief Title: Vascular Response to Isoproterenol and β2 Adrenergic Receptor Polymorphisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: yc19558-HMO-CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Isoproterenol

INTERVENTIONS:
Drug: Isoproterenol

SUMMARY:
Single nucleotide polymorphisms at codon 46 and 79 of the gene encoding for the ß2 adrenergic receptor (ß2AR) modify its pharmacological properties and may alter the response to ß2AR agonists. The goal of the present study was to evaluate the role played by the Arg16Gly and Gln27Glu polymorphisms on isoproterenol induced relaxation of internal mammary arteries segments ex-vivo.

Internal mammary leftover segments were collected from 96 patients undergoing coronary artery bypass graft operation. Four rings that were prepared from each specimen were allowed to reach equilibrium with physiological Krebs solution prior to precontraction with U46619. Using the organ bath technique, cumulative dose response curve of isoproterenol was constructed and mean EC50 calculated for each patient.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo coronary artery bypass graft operation

Exclusion Criteria:

* Chronic treatment with corticosteroids

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1999-08

PRIMARY OUTCOMES:
Mean Ec50% in response to rising concentration of isoproterenol

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Khalaila JM, Elami A, Caraco Y. Interaction between beta2 adrenergic receptor polymorphisms determines the extent of isoproterenol-induced vasodilatation ex vivo. Pharmacogenet Genomics. 2007 Oct;17(10):803-11. doi: 10.1097/FPC.0b013e3281eb8f07. PMID 17885618